CLINICAL TRIAL: NCT03887767
Title: Prognostic Value of sST2 in Cardiac Surgery on Long Term Morbimortality
Brief Title: sST2 and Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0094
Record Dates: First submitted 2019-03-05; First posted 2019-03-25 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the prognosis value of sST2 dosed before cardiac surgery on prognosis of long terme prognosis after cardiac surgery.

The patients where initialy recruted for another cohort named micro-SIRS and inflammation but the gaved their consent to analyse the blood samples for other studies

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80
* cardiac surgery includind coronary arterial bypass of valvular surgery

Exclusion Criteria:

* other surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included before cardiac surgery
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 1 year
  1 year mortality rate

SECONDARY OUTCOMES:
Number of rehospitalisation | 1 day
  Number of rehospitalisation
Number of cardiac events | 1 day
  Number of cardiac events
Number of cardiac stroke | 1 day
  Number of cardiac stroke

CONTACTS AND LOCATIONS:
Overall Officials: Kada KLOUCHE, MD PhD, Study Director — Hopital de Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC